CLINICAL TRIAL: NCT02307617
Title: Glutamate Probes in Adolescent Depression
Acronym: GPII
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paul E. Croarkin, Principal Investigator, Mayo Clinic
Other Study IDs: 14-004662
Record Dates: First submitted 2014-09-08; First posted 2014-12-04 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Major Depressive Disorder; Major Depressive Disorder, Recurrent; Major Depressive Disorder, Remitted
Keywords: Major depressive disorder; MDD; healthy control; selective serotonin reuptake inhibitor; SSRI; depression; transcranial magnetic stimulation; TMS; magnetic resonance spectroscopy; MRS; adolescent; mild MDD; mild depression; cortical excitability; cortical inhibition; cortical silent period; motor threshold; intracortical facilitation; intracortical inhibition; motor cortex; dorsolateral prefrontal cortex; DLPFC; thumb twitch; gamma aminobutyric acid; GABA; glutamate; single pulse; paired pulse
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 2: Adolescent participants who plan to start selective serotonin reuptake inhibitor (SSRI) treatment for their depression. Data will be collected prior to the start of the medication and again 6 weeks after the start of the medication.
- Medication Responders: Adolescent participants who have responded to SSRI treatment for their depression.
- Medication Non-Responders: Adolescent participants with depression that has not responded to SSRI treatment.
- Healthy Controls: Adolescent participants who have no current or past mental health diagnoses.

SUMMARY:
The purpose of this study is to learn if measures of brain chemicals from a brain scan called Magnetic Resonance Imaging and Spectroscopy (MRI/MRS) and brain activity (known as cortical excitability and inhibition) collected by Transcranial Magnetic Stimulation (TMS) are different in adolescents with depression who are in different stages of treatment.

Researchers are conducting this study to learn more about how the brain works in adolescents with depression and without depression (healthy controls). This is important because it may identify a biological marker (a measure of how bad an illness is) for depression that could one day be used to identify depressed adolescents who would benefit from certain treatments (medications for example) or to monitor how well treatments are working.

DETAILED DESCRIPTION:
This is a cross-sectional and longitudinal neurophysiology research study of 200 adolescent subjects in varying stages of major depressive disorder (MDD). The aims of this study are designed to gain an understanding of (1) the role of glutamate in the neurophysiology and pharmacologic treatment of child and adolescent MDD; (2) the role of gamma-aminobutyric acid (GABA) in the neurophysiology and pharmacologic treatment of child and adolescent MDD; (3) the trajectory of glutamatergic and GABAergic functioning in human development with MDD.

Glutamate concentrations in the anterior cingulate cortex (ACC) and left dorsolateral prefrontal (L-DLPFC) cortex will be evaluated using proton magnetic resonance spectroscopy (MRS) at 3 Tesla (3T). Glutamatergic cortical excitability measures (with motor threshold and intracortical facilitation paradigms), and GABAergic cortical inhibitory measures (with cortical silent period and intracortical inhibition paradigms) will be studied using single and paired-pulse transcranial magnetic stimulation (TMS) paradigms.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents from the ages of 13 to 21, male or female.
2. Subjects with MDD (Groups 2, 3 & 4):

   * Must have a diagnosis of Major Depressive Disorder (MDD)
   * Single episode or recurrent; moderate to severe.
   * The MDD diagnosis is based on the Kiddie Schedule for Affective Disorders and Schizophrenia for School Aged Children - Past and Lifetime (K-SADS-PL).
   * This semi-structured psychiatric interview will be administered by a psychiatrist, Ph.D. level psychologist, or equivalent professional with extensive clinical experience.
   * Must have a Childhood Depression Rating Scale-Revised (CDRS-R) score of ≥ 40
   * Must have a Clinical Global Impression Severity (CGI-S) Scale of ≥ 4
3. Group 1: (Healthy Controls; 50 Subjects): Healthy volunteers who are 13-21 years of age with no current or lifetime mental health diagnoses and no current or lifetime psychotropic medication treatment.
4. Group 2: (50 subjects): Subjects with moderate to severe MDD for which an SSRI has been clinically indicated.

   * If initiating SSRI treatment, medication must be started ± 7 days of the baseline visit
   * Subjects and parents in group 2 will be eligible to return in 6-8 weeks for a follow up visit that includes mood assessments and evaluations.
   * Subjects who have been adherent to their clinically prescribed medication will be eligible for a second MRI/MRS scan and TMS measures within 7 days of the second visit.
   * Subjects who choose not to initiate treatment with an SSRI will have a baseline visit only
   * Subjects who discontinue or change their medication after the baseline will not be eligible for a follow-up visit

   Group 3: (50 subjects): Subjects with moderate to severe MDD that has responded to treatment with an SSRI.

   • Response will be defined as a 1 (very much) or 2 (much) improved on a CGI-Improvement Scale. This is the current acceptable standard in child and adolescent psychopharmacological research.

   Group 4: (50 subjects): Subjects with moderate to severe MDD that has not responded to treatment with an SSRI as defined above with CGI scale score.
5. Subject and parent or guardian (if under age 18) must be capable of providing informed consent
6. Subjects and at least 1 parent must be fluent in English. • Subjects 18 years of age or older do not require an English-speaking parent

Exclusion Criteria:

4.2 Exclusion Criteria For all Subjects:

1. Contraindications to MRI/MRS, as determined by the MRI safety screen and MRI safety codes.
2. Subjects who are judged by the Principal Investigator to be at imminent risk for self-harm or suicide as indicated by interview or C-SSRS.
3. Pregnancy or suspected pregnancy in females.
4. Metal in the head (except the mouth*), implanted medication pumps, cardiac pacemaker (*subjects with braces will be excluded from MRI/MRS portion of the study only)
5. Prior brain surgery.
6. Risk for increased intracranial pressure such as a brain tumor.
7. Any unstable medical condition.

4.2.1 Exclusion Criteria for Healthy Control Group only:

1. Current or past mental health diagnoses in subjects or first degree relatives of subjects.
2. Current or past mental health medications.

4.2.2 Exclusion Criteria for MDD Groups only:

1. Primary Axis I or II disorder other than MDD.
2. Unprovoked seizure history, seizure disorder, history of febrile seizures, first degree relative with epilepsy
3. Taking medication(s) that lower seizure threshold
4. Any significant findings on the TMS adult safety screen (TASS).

4.2.3 Exclusion Criteria for Group 2 only:

1. Subject has started SSRI medication more than 7 days prior to the baseline visit.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This protocol will plan to screen depressed children and adolescents who are seeking treatment at Mayo Clinic in Rochester, MN, using strict inclusion and exclusion criteria. These adolescents will represent gender and minority distribution consistent with the Rochester metro/rural area demographic distribution. This study will be inclusive of all races, genders, and socioeconomic classes.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2017-04-17 (Actual)

PRIMARY OUTCOMES:
Concentrations of GABA and glutamate in the brains of adolescents with MDD. | Baseline
  Glutamate concentrations in the anterior cingulate cortex (ACC) and left dorsolateral prefrontal (L-DLPFC) cortex will be evaluated using proton magnetic resonance spectroscopy (MRS) at 3T. Glutamatergic cortical excitability measures (with motor threshold and intracortical facilitation paradigms), and GABAergic cortical inhibitory measures (with cortical silent period and intracortical inhibition paradigms) will be studied using single and paired-pulse transcranial magnetic stimulation (TMS) paradigms.
The change of GABA and glutamate concentrations in adolescents with MDD after 6 weeks of SSRI treatment. | Baseline to 6 weeks (group 2)
  Glutamate concentrations in the anterior cingulate cortex (ACC) and left dorsolateral prefrontal (L-DLPFC) cortex will be evaluated using proton magnetic resonance spectroscopy (MRS) at 3T. Glutamatergic cortical excitability measures (with motor threshold and intracortical facilitation paradigms), and GABAergic cortical inhibitory measures (with cortical silent period and intracortical inhibition paradigms) will be studied using single and paired-pulse transcranial magnetic stimulation (TMS) paradigms.

SECONDARY OUTCOMES:
The effect of glutamatergic and GABAergic functioning on human development in adolescents with MDD | Baseline
  Glutamatergic and GABAergic function will be measured using single and paired-pulse Transcranial Magnetic Stimulation (TMS) measures of cortical excitability (motor threshold and intracortical facilitation) and inhibition (cortical silent period and intracortical inhibition).
The effect of glutamatergic and GABAergic functioning on human development in adolescents with MDD after 6 weeks of SSRI treatment. | Baseline to 6 weeks (group 2)
  Glutamatergic and GABAergic function will be measured using single and paired-pulse Transcranial Magnetic Stimulation (TMS) measures of cortical excitability (motor threshold and intracortical facilitation) and inhibition (cortical silent period and intracortical inhibition).

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Croarkin, D.O., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials